CLINICAL TRIAL: NCT01454947
Title: Use of Behavioral Economics to Improve Treatment of Acute Respiratory Infections (Main Study)
Acronym: BEARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jason Doctor, Associate Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1RC4AG039115-01 (NIH); 1RC4AG039115-01 (NIH)
Record Dates: First submitted 2011-08-04; First posted 2011-10-19 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Acute Respiratory Infections (ARIs)
Keywords: Antibiotics; Inappropriate Prescribing; Respiratory Tract Infections; Behavioral Research
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- SA, AJ, PC (Experimental): Participants are given all 3 interventions.
  Interventions: Behavioral: Clinical Decision Support (CDS): Accountable Justifications; Behavioral: Audit and Feedback: Peer Comparison; Behavioral: CDS Order Sets: Suggested Alternatives
- SA, AJ (Experimental): Participants receive the Suggested Alternatives and Accountable Justification interventions, but not the Peer Comparison intervention.
  Interventions: Behavioral: Clinical Decision Support (CDS): Accountable Justifications; Behavioral: CDS Order Sets: Suggested Alternatives
- SA, PC (Experimental): Participants receive the Suggested Alternative and Peer Comparison interventions, but not the Accountable Justification intervention.
  Interventions: Behavioral: Audit and Feedback: Peer Comparison; Behavioral: CDS Order Sets: Suggested Alternatives
- AJ, PC (Experimental): Participants receive the Accountable Justification and Peer Comparison interventions, but not the Suggested Alternative intervention.
  Interventions: Behavioral: Clinical Decision Support (CDS): Accountable Justifications; Behavioral: Audit and Feedback: Peer Comparison
- Peer Comparison (PC) (Experimental): Participants receive the Peer Comparison intervention, but do not receive the Suggested Alternatives or Accountable Justification interventions.
  Interventions: Behavioral: Audit and Feedback: Peer Comparison
- Suggested Alternatives (SA) (Experimental): Participants receive the Suggested Alternatives intervention, but not the Accountable Justification or Peer Comparison interventions.
  Interventions: Behavioral: CDS Order Sets: Suggested Alternatives
- Accountable Justification (AJ) (Experimental): Participants receive the Accountable Justification intervention, but do not receive the Suggested Alternatives or Peer Comparison interventions.
  Interventions: Behavioral: Clinical Decision Support (CDS): Accountable Justifications
- Education Control (No Intervention): Participants do not receive any of the 3 interventions.

INTERVENTIONS:
Behavioral: Clinical Decision Support (CDS): Accountable Justifications — Accountable Justifications triggered by discordant prescriptions that populate the electronic health record (EHR) note with provider's rationale for guideline exceptions (AJ).
  Other Names: AJ; Accountable Justification
  Arms: AJ, PC; Accountable Justification (AJ); SA, AJ; SA, AJ, PC
Behavioral: Audit and Feedback: Peer Comparison — Performance feedback that benchmarks providers' own performance to that of their peers (PC, for Peer Comparison).
  Other Names: PC; Peer Comparison
  Arms: AJ, PC; Peer Comparison (PC); SA, AJ, PC; SA, PC
Behavioral: CDS Order Sets: Suggested Alternatives — Order Sets that are triggered by EHR workflow containing exclusively guideline concordant choices (SA, for Suggested Alternatives).
  Other Names: SA; Suggested Alternatives
  Arms: SA, AJ; SA, AJ, PC; SA, PC; Suggested Alternatives (SA)

SUMMARY:
Bacteria resistant to antibiotic therapy are a major public health problem. The evolution of multi-drug resistant pathogens may be encouraged by provider prescribing behavior. Inappropriate use of antibiotics for nonbacterial infections and overuse of broad spectrum antibiotics can lead to the development of resistant strains. Though providers are adequately trained to know when antibiotics are and are not comparatively effective, this has not been sufficient to affect critical provider practices.

The intent of this study is to apply behavioral economic theory to reduce the rate of antibiotic prescriptions for acute respiratory diagnoses for which guidelines do not call for antibiotics. Specifically targeted are infections that are likely to be viral.

The objective of this study is to improve provider decisions around treatment of acute respiratory infections.

The participants are practicing attending physicians or advanced practice nurses (i.e. providers) at participating clinics who see acute respiratory infection patients. A maximum of 550 participants will be recruited for this study.

Providers consenting to participate will fill out a baseline questionnaire online. Subsequent to baseline data collection and enrollment, participating clinic sites will be randomized to the study arms, as described below.

There will be a control arm, with clinic sites randomized in a multifactorial design to up to three interventions that leverage the electronic medical record: Order Sets that are triggered by electronic health record (EHR) workflow containing exclusively guideline concordant choices (SA, for Suggested Alternatives); Accountable Justifications triggered by discordant prescriptions that populate the note with provider's rationale for guideline exceptions (AJ); and performance feedback that benchmarks providers' own performance to that of their peers (PC, for Peer Comparisons).

The outcomes of interest are antibiotic prescribing patterns, including prescribing rates and changes in prescribing rates over time.

The intervention period will be over one year, with a one-year follow up period to measure persistence of the effect after EHR features are returned to the original state and providers no longer receive email alerts.

DETAILED DESCRIPTION:
Each consented provider will be randomized to 1 of 8 cells in a factorial design with equal probability. If results of retrospective data analysis imply that design will be improved by stratification, randomization will be stratified by factors that could influence outcomes.

Data will be collected from the clinics' Enterprise Data Warehouses which store copies of data recorded in the electronic health record. Data elements from qualifying office visits will be collected from coded portions of the electronic health record.

An encounter is eligible for intervention if the patient's diagnosis is in the selected group of acute respiratory infections. The intervention EHR functions will be triggered when clinicians initiate an antibiotic prescription or enter a diagnosis for an acute respiratory infection that has a defined Order Set. If an antibiotic from a list of frequently misprescribed antibiotics is ordered and a diagnosis has not yet been entered, providers will be prompted to enter a diagnosis. If the diagnosis entered is acute nasopharyngitis; acute laryngopharyngitis/acute upper respiratory infection; acute bronchitis; bronchitis not specified as acute or chronic; or flu; the interventions will be triggered. The diagnosis-appropriate order set will pop-up for providers in the SA arm, while clinicians randomized to the AJ arm will receive an alert and be required to enter a brief statement justifying their antibiotic prescription if antibiotics are not indicated for the diagnosis entered. This note will then be added to the patient's medical record.

Clinicians randomized to the Peer Comparison condition will receive email updates about their antibiotic prescribing practices relative to other clinicians in their practice.

ELIGIBILITY:
Inclusion Criteria:

* A practicing attending physician or advanced practice nurse ("provider") at a participating clinic in 2011-2013 who sees acute respiratory infection patients.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2011-08; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason N Doctor, PhD, Principal Investigator — University of Southern California
Locations (55):
- United States (55):
  - Altamed Anaheim Lincoln, Anaheim, California
  - Altamed Anaheim West, Anaheim, California
  - Altamed Bell Clinic, Bell, California
  - Altamed Mobile Unit Primary Care, Commerce, California
  - Altamed DVL El Monte, El Monte, California
  - Altamed El Monte Clinic, El Monte, California
  - Altamed Garden Grove Harbor, Garden Grove, California
  - Altamed Huntington Beach Clinic, Huntington Beach, California
  - Altamed PACE Rugby, Huntington Park, California
  - The Children's Clinic Family Health Center at Cesar Chavez Elementary School, Long Beach, California
  - The Children's Clinic Family Health Center at Hamilton Middle School, Long Beach, California
  - The S. Mark Taper Foundation Children's Clinic Family Health Center, Long Beach, California
  - The Children's Clinic at the Long Beach Multi-Service Center for the Homeless, Long Beach, California
  - The Vasek Polak Children's Clinic Family Health Center, Long Beach, California
  - Altamed PACE Grand Plaza, Los Angeles, California
  - Altamed William Mead Homes, Los Angeles, California
  - Altamed Commerce Clinic, Los Angeles, California
  - Altamed DVL Commerce, Los Angeles, California
  - Altamed PACE Pomona, Los Angeles, California
  - Altamed Boyle Heights Clinic, Los Angeles, California
  - Altamed Estrada Courts, Los Angeles, California
  - Altamed Ramona Gardens, Los Angeles, California
  - AltaMed 1st St Boyle Heights Clinic, Los Angeles, California
  - Altamed Zonal Clinic, Los Angeles, California
  - Altamed Montebello Clinic, Montebello, California
  - Altamed El Modena Clinic, Orange, California
  - Altamed Pico Clinic, Pico Rivera, California
  - Altamed DVL Pico, Pico Rivera, California
  - Altamed Santa Ana Main, Santa Ana, California
  - Altamed Clinic For Women, Santa Ana, California
  - Altamed Santa Ana Broadway, Santa Ana, California
  - Altamed Santa Ana Central, Santa Ana, California
  - Brigham and Women's Primary Care Associates at Foxborough, Boston, Massachusetts
  - MGH Downtown, Boston, Massachusetts
  - Mass General Medial Group, Boston, Massachusetts
  - MGH Beacon Hill, Boston, Massachusetts
  - MGH Senior Health, Boston, Massachusetts
  - Women's Health Associates, Boston, Massachusetts
  - Brigham Circle Medical Associates, Boston, Massachusetts
  - Brigham Internal Medicine Associates, Boston, Massachusetts
  - Spanish Clinic, Boston, Massachusetts
  - MGH Back Bay, Boston, Massachusetts
  - Brigham and Women's Primary Care Associates of Brookline, Brookline, Massachusetts
  - MGH Charlestown HealthCare Center, Charlestown, Massachusetts
  - MGH Chelsea HealthCare Center, Chelsea, Massachusetts
  - Brigham and Women's Physician Group, Chestnut Hill, Massachusetts
  - Gretchen and Edward Fish Center for Women's Health, Chestnut Hill, Massachusetts
  - Everett Family Practice, Everett, Massachusetts
  - Brigham Primary Physicians at Faulkner, Jamaica Plain, Massachusetts
  - Brookside Community Health Center, Jamaica Plain, Massachusetts
  - Faulkner Community Physicians, Jamaica Plain, Massachusetts
  - Southern Jamaica Plain Health Center, Jamaica Plain, Massachusetts
  - Brigham and Women's Primary Care Associates of Newton Corner, Newton, Massachusetts
  - Mass General Revere HealthCare Center, Revere, Massachusetts
  - Mass General West Medical Group, Waltham, Massachusetts

REFERENCES:
- [Background] Meeker D, Linder JA, Fox CR, Friedberg MW, Persell SD, Goldstein NJ, Knight TK, Hay JW, Doctor JN. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):562-70. doi: 10.1001/jama.2016.0275. PMID 26864410
- [Derived] Doctor JN, Goldstein NJ, Fox CR, Linder JA, Persell SD, Stewart EP, Knight TK, Meeker D. Clinician Job Satisfaction After Peer Comparison Feedback: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2317379. doi: 10.1001/jamanetworkopen.2023.17379. PMID 37289454
- [Derived] Gong CL, Zangwill KM, Hay JW, Meeker D, Doctor JN. Behavioral Economics Interventions to Improve Outpatient Antibiotic Prescribing for Acute Respiratory Infections: a Cost-Effectiveness Analysis. J Gen Intern Med. 2019 Jun;34(6):846-854. doi: 10.1007/s11606-018-4467-x. Epub 2018 May 8. PMID 29740788
- [Derived] Gong CL, Hay JW, Meeker D, Doctor JN. Prescriber preferences for behavioural economics interventions to improve treatment of acute respiratory infections: a discrete choice experiment. BMJ Open. 2016 Sep 22;6(9):e012739. doi: 10.1136/bmjopen-2016-012739. PMID 27660322
- [Derived] Persell SD, Friedberg MW, Meeker D, Linder JA, Fox CR, Goldstein NJ, Shah PD, Knight TK, Doctor JN. Use of behavioral economics and social psychology to improve treatment of acute respiratory infections (BEARI): rationale and design of a cluster randomized controlled trial [1RC4AG039115-01]--study protocol and baseline practice and provider characteristics. BMC Infect Dis. 2013 Jun 27;13:290. doi: 10.1186/1471-2334-13-290. PMID 23806017

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Education Control | Suggested Alternatives (SA) | Accountable Justification (AJ) | Peer Comparison (PC) | SA, AJ | SA, PC | AJ, PC | SA, AJ, PC
Started | 27 | 42 | 35 | 20 | 34 | 35 | 27 | 28
Completed | 24 | 38 | 32 | 19 | 33 | 32 | 26 | 23
Not Completed | 3 | 4 | 3 | 1 | 1 | 3 | 1 | 5

BASELINE CHARACTERISTICS:
Population: Enrolled Clinicians
Groups:
- Total: Total of all reporting groups
Arm/Group | Education Control | Suggested Alternatives (SA) | Accountable Justification (AJ) | Peer Comparison (PC) | SA, AJ | SA, PC | AJ, PC | SA, AJ, PC | Total
Number analyzed (Participants) | 27 | 42 | 35 | 20 | 34 | 35 | 27 | 28 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (12) | 49 (10) | 49 (9) | 46 (9) | 48 (9) | 51 (11) | 48 (10) | 46 (9) | 48 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 30 | 22 | 12 | 24 | 25 | 15 | 16 | 157
  Male | 14 | 12 | 13 | 8 | 10 | 10 | 12 | 12 | 91

OUTCOME MEASURES:

1. Primary Outcome: Inappropriate Antibiotic Prescribing Rate for Qualifying Acute Respiratory Infection Diagnoses
Description: Assess inappropriate antibiotic prescribing rates (relative to all practices that did not receive the intervention) for antibiotic-inappropriate acute respiratory tract infection visits and no concomitant reason for antibiotic prescribing. based on the following non-antibiotic-appropriate International Statistical Classification of Diseases, version 9 (ICD-9) diagnoses:
  460 Acute nasopharyngitis (common cold)
  465 Acute laryngopharyngitis/acute upper respiratory infection
  466 Acute bronchitis
  490 Bronchitis not specified as acute or chronic
  487 Flu
Time Frame: 18 months
Population: We identified a total of 16,959 non-antibiotic-appropriate acute respiratory infection (ARI) visits. Visits were categorized as inappropriate if there were diagnosis codes for non-specific upper respiratory infections, acute bronchitis, and/or influenza.
Measure: Number (95% Confidence Interval); unit: proportion of visits
Units Other Than Participants: Qualifying ARI visits
Groups:
- Control: Participants received no study interventions
- Suggested Alternatives + Accountable Justification: Participants receive the Suggested Alternatives and Accountable Justification interventions, but do not receive the Peer Comparison intervention
- Suggested Alternatives + Peer Comparison: Participants receive the Suggested Alternatives and Peer Comparison interventions, but do not receive the Accountable Justification intervention
- Accountable Justification + Peer Comparison: Participants receive the Accountable Justification and Peer Comparison interventions, but do not receive the Suggested Alternatives intervention
- SA+AJ+PC: Participants receive all three interventions: Suggested Alternatives, Accountable Justification, and Peer Comparison interventions
Arm/Group | Control | Suggested Alternatives (SA) | Accountable Justification (AJ) | Peer Comparison (PC) | Suggested Alternatives + Accountable Justification | Suggested Alternatives + Peer Comparison | Accountable Justification + Peer Comparison | SA+AJ+PC
Number analyzed (Participants) | 27 | 42 | 35 | 20 | 34 | 35 | 27 | 28
Number analyzed (Qualifying ARI visits) | 2095 | 2388 | 1979 | 1620 | 2131 | 2014 | 2240 | 2492
proportion of visits | 0.20 [0.10 to 0.31] | 0.19 [0.06 to 0.66] | 0.08 [0.03 to 0.23] | 0.09 [0.03 to 0.31] | 0.07 [0.02 to 0.24] | 0.01 [0.00 to 0.08] | 0.03 [0.00 to 0.18] | 0.03 [0.00 to 0.22]

2. Secondary Outcome: Encounters Closely Following the Index Encounter for Serious Diagnoses
Description: Within intervention-qualifying acute respiratory infections (ARI) encounters where no antibiotic was prescribed, we will monitor return visit rates for the specified diagnoses and other acute respiratory infection diagnoses (ICD-9), including whooping cough (033.9), rheumatic fever (390-392) and pneumonia (481-487).
Time Frame: 18 months
Population: Overall number of units analyzed is the number of intervention-qualifying acute respiratory infections (ARI) encounters where no antibiotic was prescribed. Intervention-qualifying ARI encounters include all ARI visits eligible for the suggested alternatives and accountable justification interventions (not limited to the antibiotic-inappropriate ARI diagnoses that define the primary outcome).
Measure: Count of Units; unit: Qualifying encounters
Units Other Than Participants: Qualifying encounters
Arm/Group | Control | Suggested Alternatives (SA) | Accountable Justification (AJ) | Peer Comparison (PC) | Suggested Alternatives + Accountable Justification | Suggested Alternatives + Peer Comparison | Accountable Justification + Peer Comparison | SA+AJ+PC
Number analyzed (Participants) | 27 | 42 | 35 | 20 | 34 | 35 | 27 | 28
Number analyzed (Qualifying encounters) | 3245 | 4579 | 4622 | 3781 | 5717 | 5993 | 3398 | 4164
Qualifying encounters | 14 | 16 | 16 | 13 | 22 | 23 | 48 | 15
Statistical Analysis 1: Comparison: Control vs Suggested Alternatives (SA) vs Accountable Justification (AJ) vs Peer Comparison (PC) vs Suggested Alternatives + Accountable Justification vs Suggested Alternatives + Peer Comparison vs Accountable Justification + Peer Comparison vs SA+AJ+PC; Test type: Superiority; p = 0.007, 2 proportion Z-test — P values computed using difference between proportions (z value) with Bonferroni correction

ADVERSE EVENTS:
Time Frame: For antibiotic-inappropriate visits in which no antibiotic was prescribed, we assessed return visits within 30 days for the presence of complications potentially attributable to untreated bacterial infections
Description: Intervention-qualifying acute respiratory infections (ARI) encounters include all ARI visits eligible for the suggested alternatives and accountable justification interventions (not limited to the antibiotic-inappropriate ARI diagnoses that define the primary outcome). A Diagnosis of Concern (DoC) was based on International Classification of Diseases version 9 (ICD9) codes of concern at revisit.
Arm/Group | Education Control | Suggested Alternatives (SA) | Accountable Justification (AJ) | Peer Comparison (PC) | SA, AJ | SA, PC | AJ, PC | SA, AJ, PC
Serious Adverse Events (participants affected / at risk) | 0/3245 | 0/4579 | 0/4622 | 0/3781 | 0/5717 | 0/5993 | 0/3398 | 0/4164
Other Adverse Events (participants affected / at risk) | 14/3245 | 16/4579 | 16/4622 | 13/3781 | 22/5717 | 23/5993 | 48/3398 | 15/4164
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Education Control (N=3245) | Suggested Alternatives (SA) (N=4579) | Accountable Justification (AJ) (N=4622) | Peer Comparison (PC) (N=3781) | SA, AJ (N=5717) | SA, PC (N=5993) | AJ, PC (N=3398) | SA, AJ, PC (N=4164)
return visits for bacterial infections occurring within 30 days of study qualifying ARI visit where (Infections and infestations) | 14 | 16 | 16 | 13 | 22 | 23 | 48 | 15 — For antibiotic-inappropriate visits in which no antibiotic was prescribed, we assessed return visits within 30 days for the presence of complications potentially attributable to untreated bacterial infections

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes